CLINICAL TRIAL: NCT02411630
Title: Structural and Partnership Factors Affecting Adherence to Pre-exposure Prophylaxis (PREP)Among Young Men Who Have Sex With Men
Brief Title: Factors Affecting PrEP Adherence
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 123
Record Dates: First submitted 2014-01-23; First posted 2015-04-08 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-12

CONDITIONS: HIV Infection
Keywords: PrEP; HIV Prevention
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interactive Questionnaire System (iQS): An Interactive Questionnaire System (iQS) will be administered twice. First at study entry (ATN 110/113 week 24 visit) and second at week 24 (ATN 110/113 week 48 visit). The questionnaire will assess adherence as well as how structural (physical settings) and partnership factors affect adherence of YMSM to PrEP with FTC/TDF (Truvada®).
  Interventions: Drug: Emtricitabine/tenofovir disoproxil

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil — ATN 123 participants will not be administered Emtricitabine /Tenofovir disoproxil fumarate (Truvada®) as part of the ATN 123 study, but as part of the parent studies, ATN 110 or ATN 113. In order to be eligible for ATN 123, all participants must be co-enrolled in ATN 110 or ATN 113.
  The only intervention for ATN 123 is the administration of the Interactive Questionnaire System (iQS), which is a new method to collect data on adherence. It will be utilized to collect adherence data across a variety of devices (i.e., computer/laptop, smartphone, tablet, etc.). Accuracy of this method will be determined; preference for this mode of data collection compared to other methods for adherence reporting used in the parent studies will be assessed.
  Other Names: Truvada®; FTC/TFV

SUMMARY:
The purpose of this study is to test a new way to take a questionnaire that asks about adherence (whether the person is taking the medicine correctly). This new questionnaire is called Interactive Questionnaire System (iQS). In this study, the iQS will be tested on HIV-negative young men who have sex with men (YMSM) who are taking PrEP as part of another study, either ATN 110 or ATN 113.

DETAILED DESCRIPTION:
Among Men who have Sex with Men (MSM) in the U.S., Human Immunodeficiency Virus (HIV) incidence has remained highest in those less than 30 years of age, demonstrating the need for new ways to prevent HIV in Young Men who have Sex with Men (YMSM). Pre-exposure Prophylaxis or PrEP is the use of a daily medication to prevent HIV infection. In order for PrEP to work the pills must be taken, so adherence is a very important part of PrEP. Efforts to accurately assess adherence to PrEP have been hindered because participants do not always accurately report adherence and the flawed methods that have been used to measure adherence. In previous studies it has been shown that participants over-report adherence when compared to drug concentration levels in blood. Although drug-levels can be used to monitor adherence, the cost can be prohibitive and specimens may be difficult to collect in real-time. This means that better and more accurate assessments of PrEP adherence from self-reports are needed in order for PrEP to achieve wide-spread use.

This longitudinal pilot sub-study of ATN 110 and ATN 113 (Project PrEPare - An Open Label Demonstration Project and Phase II Safety Study of Pre-Exposure Prophylaxis Use Among Young Men Who Have Sex With Men (YMSM) in the United States) aims to assess how structural (physical settings) and partnership factors affect adherence of YMSM to PrEP. This study will compare levels of adherence reported in the Interactive Questionnaire System (iQS) to those collected in ATN 110 or ATN 113 by Audio Computer Assisted Self Interview (ACASI), Wisepill, and drug concentration levels in blood and hair. The iQS will be administered at study entry and week 24 visits. PrEP, Emtricitabine/Tenofovir disoproxil fumarate (Truvada®), will be administered as part of the ATN 110 and ATN 113 protocols. Study drug will not be administered as part of this study, ATN 123.

ELIGIBILITY:
Inclusion Criteria:

* Concurrent enrollment in ATN 110 or ATN 113 and prescribed FTC/TDF (Emtricitabine/Tenofovir disoproxil fumarate (Truvada®)) for PrEP;
* Ability to understand written and spoken English; and
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Appears visibly distraught or presence of active serious psychiatric symptoms (e.g., active hallucinations, suicidal, homicidal, or exhibiting violent behavior) at the time of consent; and
* Intoxicated or under the influence of alcohol or other substances at the time of consent.

Ages: 15 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants in this study will be HIV-1 uninfected YMSM, including transgender women, ages 15 through 22 years, inclusive at the time of consent into the parent protocol, currently enrolled in ATN 110 or ATN 113 and prescribed FTC/TDF (Truvada®) for PrEP.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Missing Data in the Interactive Questionnaire System (iQS) questionnaire | Week 0
  To assess preference of the iQS as a way to measure adherence to Pre-Exposure Prophylaxis (PrEP) in PrEP clinical trials, completion rates; pattern of skipped or incomplete responses by variables will be analyzed.
Number of Missing Data in the Interactive Questionnaire System (iQS) questionnaire | Week 24
  To assess preference of the iQS as a way to measure adherence to Pre-Exposure Prophylaxis (PrEP) in PrEP clinical trials, completion rates; pattern of skipped or incomplete responses by variables will be analyzed.
Preference for Interactive Questionnaire System (iQS) compared to Audio Computer Assisted Self Interview (ACASI) or Wisepill | Week 0
  Preference for the iQS method compared to the ACASI and Wisepill will be assessed as reported by participants.
Preference for Interactive Questionnaire System (iQS) compared to Audio Computer Assisted Self Interview (ACASI) or Wisepill | Week 24
  Preference for the iQS method compared to the ACASI and Wisepill will be assessed as reported by participants.
Adherence to Pre-Exposure Prophylaxis (PrEP) Reports by Mode: Interactive Questionnaire System (iQS) vs. Wisepill vs. Audio Computer Assisted Self Interview (ACASI) | Week 0
  Self reports in iQS, Wisepill, and ACASI will be compared to measured drug concentration levels in blood and hair. The iQS is administered as part of this study (ATN 123). The ACASI, Wisepill and drug concentration levels in blood and hair are collected as part of the parent studies (ATN 110 or ATN 113)
Adherence to Pre-Exposure Prophylaxis (PrEP)Reports by Mode: Interactive Questionnaire System (iQS) vs. Wisepill vs. Audio Computer Assisted Self Interview (ACASI) | Week 24
  Self reports in iQS, Wisepill, and ACASI will be compared to measured drug concentration levels in blood and hair. The iQS is administered as part of this study (ATN 123). The ACASI, Wisepill and drug concentration levels in blood and hair are collected as part of the parent studies (ATN 110 or ATN 113)

OTHER OUTCOMES:
Association of components of the Person Environment Theoretical Framework (PETF) (specifically physical setting (structural) and social climate (partnership factors)) with adherence to PrEP among YMSM | Week 0 and Week 24
  Components of Person Environment Theoretical Framework (PETF), specifically physical setting (structural) and social climate (partnership factors)) and adherence change over time will be assessed by comparing reports between the first administration of the iQS at Week 0 and the second administration at week 24.
Association of components of the PETF (physical setting (structural) and social climate (partnership factors)) with change over time. | Week 0 and Week 24
  To assess how components of the PETF (physical setting (structural) and social climate (partnership factors)) change over time by comparing reports between the first administration of the iQS at Week 0 and the second administration at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Pamina M Gorbach, MHS, DrPH, Study Chair — University of California, Los Angeles; Michelle Lally, MD, MSc, Study Chair — Alpert Medical School, Brown University
Locations (12):
- United States (12):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Children's Hospital of Denver, Aurora, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University-Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas